CLINICAL TRIAL: NCT04266574
Title: BRAIN-targeted Goal-directed Therapy in High-risk Patients undeRgOing Major electIve SurgEry: the BRAIN-PROMISE Study
Acronym: BRAINPROMISE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1211
Record Dates: First submitted 2020-02-10; First posted 2020-02-12 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Surgery; Perioperative Complication
MeSH Terms: interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Near Infrared Spectroscopy (NIRS) (Experimental)
  Interventions: Device: Near Infrared Spectroscopy (NIRS)
- Standard Care (Active Comparator)
  Interventions: Device: Standard Care

INTERVENTIONS:
Device: Near Infrared Spectroscopy (NIRS) — The anesthesiologist will apply optodes before induction of anesthesia and before preoxygenation, to detect baseline NIRS level, NIRS will be monitored continuously up to post-anaesthesia care unit (PACU) discharge, or up to three the investigator's after ICU admission.
  When a decrease in NIRS value over 10% is detected, or if NIRS value is below 60%, patients will start hemodynamic optimization, to reverse the reduction in NIRS and return to baseline values, according to a predefined protocol.
  Arms: Near Infrared Spectroscopy (NIRS)
Device: Standard Care — Controls will be treated according to standard of care, maintaining a MAP≥65 and an adequate cardiac output according to the hemodynamic monitoring chosen by the anesthesiologist (invasive blood pressure monitoring or pulse contour monitors). NIRS will be recorded also in controls, but caring anesthesiologists will be blinded to NIRS.
  Arms: Standard Care

SUMMARY:
The aim of the study is to further understand whether the use of non-invasive monitoring NIRS (Near Infrared Spectroscopy) is useful in reducing postoperative complications in high-risk patients undergoing elective surgery.

DETAILED DESCRIPTION:
Background:

Perioperative complications lead to impaired quality of life as well as prolonged disability. In high risk patients, early hemodynamic optimization with the goal of achieving and maintaining tissue oxygenation in the perioperative period has resulted in an improvement of outcomes and a reduction in surgery-related complications. Maintenance of adequate oxygen delivery to tissue, is one of the fundamental aspects of anesthesia. Regional Oxygen Saturation of the brain tissue (rSO2) as measured by near-infrared spectroscopy (NIRS) is a promising tool in vascular surgery and cardiac surgery for the monitoring of global cerebral perfusion.

Objectives:

This study has the purpose to assess whether an rSO2-based hemodynamic optimization algorithm is able to reduce overall perioperative complications in high risk patients.

Design:

BRAIN-PROMISE is a monocentric, randomized controlled trial.

Population:

Hypertensive elderly or frail patients undergoing major surgery.

Experimental Intervention:

Cases will be managed using a NIRS-targeted goal directed therapy.

Control Intervention:

Controls will be managed according to standard care.

Outcomes:

The primary outcome are the incidence of perioperative complications at 30 days and the percentage of successful reversal of reduction in NIRS.

Trial size:

A total of 200 patients will be randomized.

ELIGIBILITY:
Inclusion Criteria:

* hypertensive patients with American Society of Anesthesiologists (ASA) score≥ 2 with either Age ≥ 65 years or frailty score ≥5
* presence of an arterial catheter during anesthesia
* planned high-risk surgery (abdominal, vascular, urologic, thoracic one-lung ventilation (OLV) procedures), longer than 60 minutes, in general anesthesia
* ability to give informed consent according to International Conference on Harmonization ICH/ Good Clinical Practice (GCP), and national/local regulations

Exclusion Criteria:

* Unable to consent to study inclusion
* Language barrier
* Severe neurological or psychiatric disease
* End-stage dementia
* Total Intravenous anesthesia
* No use of hypertensive medication at home.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-11-17 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
The overall incidence of perioperative complications (including postoperative cognitive dysfunction and delirium). | 30 day after randomization
Percentage of successful reversal of reduction in NIRS, according to the hemodynamic optimization protocol. | intraoperative

SECONDARY OUTCOMES:
NIRS variations over time, and according to interventions | intraoperative
Percentage of time with NIRS within safety limits (<10% reduction) | intraoperative
Bispectral index (BIS) over time | intraoperative
Mean arterial pressure (MAP) over time | intraoperative
sevorane concentration over time | intraoperative
Use of vasopressors and fluids to maintain MAP | intraoperative
Evaluate fluid administration | intraoperative

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Cecconi, Prof, MD, Principal Investigator — Humanitas Research Hospital IRCCS, Rozzano-Milan
Locations (1):
- Humanitas Research Hospital, Rozzano, Milan, Italy

REFERENCES:
- [Derived] Greco M, Calgaro G, Cavallo M, Pugliese S, Mascari M, Piccirillo F, Pradella A, Piccioni F, Cecconi M. Brain-targeted goal-directed therapy in high-risk patients undergoing major elective surgery: Study protocol for the BRAIN-PROMISE randomized trial. Contemp Clin Trials. 2025 Jul;154:107940. doi: 10.1016/j.cct.2025.107940. Epub 2025 May 4. PMID 40328360